CLINICAL TRIAL: NCT04508790
Title: A Phase 2 Trial of Leflunomide, Pomalidomide, and Dexamethasone for Relapsed/Refractory Multiple Myeloma
Brief Title: Leflunomide, Pomalidomide, and Dexamethasone for the Treatment of Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19418; NCI-2020-01962 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19418 (Other: City of Hope Medical Center)
Record Dates: First submitted 2020-04-23; First posted 2020-08-11 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Leflunomide; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (leflunomide, pomalidomide, dexamethasone) (Experimental): Patients receive leflunomide PO on days 1-28, pomalidomide PO on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Drug: Leflunomide; Drug: Pomalidomide

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Leflunomide — Given PO
  Other Names: Arava; SU101
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC-4047; Imnovid; Pomalyst

SUMMARY:
This phase II trial studies how well leflunomide, pomalidomide, and dexamethasone work for the treatment of multiple myeloma that has come back (relapsed) or does not respond to treatment (refractory). Leflunomide may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Immunotherapy with pomalidomide, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving leflunomide with pomalidomide and dexamethasone may work better in treating multiple myeloma compared to pomalidomide and dexamethasone alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the response rate and to evaluate the antitumor activity of the three-drug combination, leflunomide, pomalidomide, and dexamethasone, in patients with relapsed/refractory multiple myeloma.

SECONDARY OBJECTIVES:

I. To characterize and evaluate toxicities, including type, frequency, severity, attribution, time course, and duration.

II. To obtain estimates of response duration, depth of response, clinical benefit, and survival (overall and progression-free).

OUTLINE:

Patients receive leflunomide orally (PO) on days 1-28, pomalidomide PO on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Life expectancy > 3 months
* Diagnosis of multiple myeloma with measurable disease as defined by:

  * M-protein quantities >= 0.5 g/dL by serum protein electrophoresis (sPEP) or
  * >= 200 mg/24 hour urine collection by urine protein electrophoresis (uPEP) or
  * Serum free light chain (FLC) > 10.0 mg/dL involved light chain and an abnormal kappa/lambda ration in subjects without detectable serum or urine M-protein or
  * For subjects with immunoglobulin class A (IgA) myeloma whose disease can only be reliably measured by quantitative immunoglobulin measurement, a serum IgA level >= 0.50 g/dL
* Relapsed or refractory to at least 1 prior line of therapy, including both a proteasome inhibitor and an immunomodulatory drug, and for whom transplant is not recommended. Participants may opt for a delayed transplant at a later time, if appropriate
* Fully recovered from the acute toxic effects (except alopecia) to =< grade 2 to prior anti-cancer therapy
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L (performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)

  * NOTE: Screening ANC should be independent of granulocyte- and granulocyte/macrophage colony stimulating factor (G-CSF and GM-CSF) support for at least 1 week and of pegylated G-CSF for at least 2 weeks
* Platelets >= 75.0 x 10^9/L (performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)

  * NOTE: Screening platelet count should be independent of platelet transfusions for at least 2 weeks
* Hemoglobin >= 8.0 g/dL (performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)

  * NOTE: Transfusion support is allowed
* Total bilirubin =< 2 X upper limit of normal (ULN) (unless has Gilbert's disease) (performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Aspartate aminotransferase (AST) =< 3.5 x ULN (performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Alanine aminotransferase (ALT) =< 3.5 x ULN (performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Alkaline phosphatase < 5 x ULN (performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Creatinine clearance of >= 30 mL/min per 24 hour urine test (performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 4 weeks after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Prior treatment with leflunomide
* Patients who are pomalidomide refractory, defined as subjects who progress on or within 60 days of pomalidomide when given as a single agent or in combinatorial therapies. Prior exposure to pomalidomide without refractoriness is allowed
* Current or planned use of other anti-myeloma therapies besides leflunomide, pomalidomide, and dexamethasone
* Current or planned growth factor or transfusion support until after initiation of treatment
* Prior allogeneic transplant
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents
* Positive for tuberculosis or latent tuberculosis (TB)
* Positive for hepatitis A, B, or C
* Known human immunodeficiency virus (HIV) infection
* Prior diagnosis of rheumatoid arthritis
* Acute active infection requiring systemic therapy within 2 weeks prior to enrollment
* Subject has history of anaphylaxis to thalidomide, lenalidomide, pomalidomide, cholestyramine or dexamethasone
* Non-hematologic malignancies within the past 3 years, with the exceptions of

  * Adequately treated basal cell or squamous cell skin cancer,
  * Carcinoma in situ of the cervix,
  * Prostate cancer < Gleason grade 6 with stable prostate specific antigen (PSA), or
  * Successfully treated in situ carcinoma of the breast
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2027-02-14 (Estimated); Study Completion 2027-02-14 (Estimated)

PRIMARY OUTCOMES:
Overall response | Up to 1 year
  Clopper Pearson binomial 95% confidence intervals will be calculated.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days after last dose
  Graded according to Common Terminology Criteria for Adverse Events (CTCAE) version (v)5. Observed toxicities will be summarized, for all dose levels, in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.
Response duration | Up to 1 year
  Will be estimated using the product-limit method of Kaplan and Meier.
Depth of response | Up to 1 year
  Will be estimated using the product-limit method of Kaplan and Meier.
Clinical benefit response | Up to 1 year
  Clopper Pearson binomial 95% confidence intervals will be calculated.
Overall survival | Up to 1 year
  Will be estimated using the product-limit method of Kaplan and Meier.
Minimal residual disease (MRD) status | Up to 1 year
  A patient will be considered as having minimal residual diseases if a positive result is obtained using the Adaptive MRD testing. MRD testing will be performed at Adaptive Biotechnologies.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Rosenzweig, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States